CLINICAL TRIAL: NCT04723823
Title: Mapping of Motor and Sensory Brain Activity Using fMRI
Brief Title: Sensorimotor Imaging for Brain-Computer Interfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Carnegie Mellon University (Other); Synchron Medical, Inc. (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jennifer Collinger, PhD, Associate Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19060314; 1UG3NS120191-01 (NIH)
Record Dates: First submitted 2021-01-07; First posted 2021-01-26 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Functional Neuroimaging
Keywords: tetraplegia; ALS; amyotropic lateral sclerosis
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Intervention Model Description: Participants will be asked to imagine movements or sensensations while brain activity is measured with fMRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with spinal cord injury (SCI) (Experimental): Individuals will be asked to imagine movements or sensations while fMRI is used to measure brain activity.
  Interventions: Other: Motor or sensory imagery with fMRI
- Individuals with amotrophic lateral sclerosis (ALS) (Experimental): Individuals will be asked to imagine movements or sensations while fMRI is used to measure brain activity.
  Interventions: Other: Motor or sensory imagery with fMRI

INTERVENTIONS:
Other: Motor or sensory imagery with fMRI — Brain activity will be measured using fMRI while participants imagine different movements or sensations in order to assess the organization of sensorimotor cortical activity after injury

SUMMARY:
The investigators will use fMRI to map movement activity in motor and somatosensory cortex using enriched imagery in people with chronic tetraplegia. The investigators expect that somatotopic organization of movement activity will be preserved in people with upper limb impairments, which can be quantified using the strength, area, and location of sensorimotor activity. Accurate mapping of the motor and somatosensory cortices using covert stimuli will help guide brain-computer interface (BCI) electrode design and placement. Moreover, these advanced mapping procedures will provide new insights into the functional interactions between sensory and motor areas of the brain after injury or disease.

DETAILED DESCRIPTION:
BACKGROUND: Advanced understanding of brain structure and function has improved the diagnosis and treatment of neurological disorders such as epilepsy, stroke, and spinal cord injury (SCI). Over half a century ago, the pioneering studies of Penfield used electrical stimulation of motor and sensory areas of cerebral cortex and revealed a distinct somatotopic organization of the brain. Today, this and additional knowledge of neuronal coding functions are being used to develop revolutionary devices that interface directly with motor and sensory neurons in the brain to establish functional connections with prosthetic and assistive devices. These so-called brain-computer interfaces (BCIs) require electrodes to be placed precisely in brain areas responsible for volitional control and sensation of limb movements, particularly the arm and hand regions. Mapping those brain regions is possible using functional magnetic resonance imaging (fMRI). However, such mapping studies are difficult to perform in persons with motor and sensory impairments. People with ALS and SCI have disrupted efferent and afferent pathways between the cortex and the limbs making it necessary to rely on covert techniques, such as kinesthetic motor imagery, to map sensorimotor brain activity in order to guide BCI electrode placement or to study cortical plasticity resulting from injury or intervention. Challenges associated with brain mapping after injury likely contribute to the widely varying reports regarding the extent and prevalence of functional reorganization occurring in the brain following SCI. fMRI is a non-invasive tool that allows for measurement of motor and sensory-related brain activity with minimal risk to study participants.

SIGNIFICANCE: Restoration of upper limb function is a top priority for individuals with tetraplegia. It is estimated that 236,000-327,000 people in the United States have a spinal cord injury. Approximately 17% of people with SCI have high tetraplegia (injury at cervical levels C1-C4) although this percentage has been increasing in recent years. People with high tetraplegia are the most likely group to benefit from BCI-controlled neuroprosthetics, although the covert mapping strategies developed in this proposal could be used to study sensorimotor activation and plasticity in anyone with motor or sensory impairment including amputation. Sophisticated, motorized prostheses are being developed that enable natural upper limb movement and have advanced sensing capabilities. People with tetraplegia would like to restore function to their own limbs using FES, but this technology needs further advancement and does not replace sensation, which may still require a BCI. While FES research and development continues, people with tetraplegia could take advantage of motorized prostheses by mounting them to their wheelchair. Motorized prostheses can provide function comparable to that of an intact limb, but a high degree-of-freedom control interface is needed and BCI is one possible solution.

Functional neuroimaging can be used to guide BCI electrode placement in order to tap into existing sensorimotor circuits. Imagery-based brain mapping also enables the study of cortical plasticity which could be useful for understanding maladaptive cortical changes that occur after injury or beneficial changes resulting from rehabilitation interventions. Just as pre-surgical brain mapping may help identify individuals who are best suited for a BCI, covert brain mapping in someone with motor and sensory impairments may inform the type of rehabilitation paradigm that is most likely to have a benefit. The potential benefit of being able to study cortical plasticity in the absence of movement or sensation is wide-reaching as it could be applied to patients with SCI, amputation, stroke, neurodegenerative diseases like amyotrophic lateral sclerosis, or other sensorimotor impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Normal or corrected to normal vision
3. Impairment of at least one arm/hand as a result of cervical spinal cord injury or amyotrophic lateral sclerosis. The ALS diagnosis should be possible, probable, or definite ALS based on El Escorial criteria.
4. Decreased or absent sensation or impaired hand movement
5. Score of <10 on the Short Blessed Test cognitive assessment

Exclusion Criteria:

1. Pacemaker, baclofen pump, cochlear implant or other electronic implanted device
2. Metallic implant that is unsafe for 3T MRI
3. Pregnant females
4. Individuals who weigh over 300 pounds (because of MRI risks/space)
5. Individuals who have difficulty breathing when laying down (orthopnea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Collinger, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We may share coded imaging data with other researchers.
Supporting Information: ICF
Time Frame: Deidentified data will be shared upon request to the PI and completion of a data sharing agreement.
Access Criteria: People can submit a request to download the data. Requests will be approved after completion of a brief data use agreement. The study PI will review requests to ensure that they are intended for academic purposes.
URL: https://doi.org/10.18120/0vfn-hm81

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 individuals with spinal cord injury: recruited from University of Pittsburgh Physical Medicine & Rehabilitation research registry.
  3 individuals with amyotrophic lateral sclerosis: recruited from University of Pittsburgh/UPMC neurologist, David Lacomis, MD.
Pre-assignment Details: All individuals were safety screened and underwent functional magnetic resonance imaging. No individuals were excluded.
Groups:
- S1/ SCI Participants: fMRI w/ Motor or Sensory Imagery: Individuals will be asked to attempt finger and hand movements while fMRI is used to measure brain activity.
  Motor or sensory imagery: Brain activity will be measured using fMRI while participants imagine different movements or sensations in order to assess the organization of sensorimotor cortical activity after injury.
- M1/ ALS: fMRI w/ Motor or Sensory Imagery: Individuals will be asked to attempt ankle, knee, toe, and hand movements while fMRI is used to measure brain activity.
  Motor or sensory imagery: Brain activity will be measured using fMRI while participants imagine different movements or sensations in order to assess the organization of sensorimotor cortical activity.
Period: Overall Study
Arm/Group | S1/ SCI Participants: fMRI w/ Motor or Sensory Imagery | M1/ ALS: fMRI w/ Motor or Sensory Imagery
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Individuals were pre-screened over the phone using an IRB-approved phone screening script. Individuals answered yes or no to certain eligibility criteria.
Groups:
- Participants With Spinal Cord Injury: Individuals will be asked to imagine movements or sensations while fMRI is used to measure brain activity.
  Sensory imagery: Brain activity will be measured using fMRI while participants imagine different movements or sensations in order to assess the organization of sensorimotor cortical activity after injury
- Participants With Amyotrophic Lateral Sclerosis: Individuals will be asked to imagine movements or sensations while fMRI is used to measure brain activity.
  Motor imagery: Brain activity will be measured using fMRI while participants imagine different movements or sensations in order to assess the organization of sensorimotor cortical activity after injury
- Total: Total of all reporting groups
Arm/Group | Participants With Spinal Cord Injury | Participants With Amyotrophic Lateral Sclerosis | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Full Range); unit: years] | 68.33 [60 to 76] | 26 [18 to 32] | 41.88 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8
Participants with movement-related brain activation [Count of Participants; unit: Participants] — Number of individuals who showed movement-related brain activity.
  Participants | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Peak Activity Volume: Right D1 Attempt Movement Activity at S1 - SCI
Description: Volume of peak activity strength in sensorimotor cortex for attempted movement of right thumb (D1).
Time Frame: Single visit
Population: Individuals with hand impairment due to cervical spinal cord injury
Measure: Mean (Full Range); unit: mm^3
Groups:
- Individuals With SCI: Individuals with arm/hand impairment due to SCI
Arm/Group | Individuals With SCI
Number analyzed (Participants) | 5
mm^3 | 893.6 [66 to 3355]

2. Primary Outcome: Peak Activity Volume: Right D2 Attempt Movement Activity at S1 - SCI
Description: Volume of primary activation within sensorimotor cortex for attempted movement of the right index finger (D2)
Time Frame: Single visit
Population: Individuals with hand impairment due to cervical spinal cord injury
Measure: Mean (Full Range); unit: mm^3 (cubic millimeters)
Groups:
- Individuals With Spinal Cord Injury: Individuals with hand impairment due to spinal cord injury
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 5
mm^3 (cubic millimeters) | 549 [138 to 1038]

3. Primary Outcome: Peak Activity Volume: Right D3 Attempt Movement Activity at S1 - SCI
Description: Volume of primary activation within sensorimotor cortex for attempted movement of the right middle finger (D3)
Time Frame: Single visit
Population: Individuals with hand impairment due to cervical spinal cord injury
Measure: Mean (Full Range); unit: mm^3 (cubic millimeters)
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 5
mm^3 (cubic millimeters) | 391.75 [41 to 790]

4. Primary Outcome: Peak Activity Volume: Right D4 Attempt Movement Activity at S1 - SCI
Description: Volume of primary activation within sensorimotor cortex for attempted movement of the right ring finger (D4)
Time Frame: Single visit
Population: Individuals with hand impairment due to cervical spinal cord injury
Measure: Mean (Full Range); unit: mm^3 (cubic millimeters)
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 5
mm^3 (cubic millimeters) | 221.5 [36 to 397]

5. Primary Outcome: Peak Activity Volume: Right Hand Grasp Overt/Attempt Movement Activity at S1 - SCI
Description: Volume of peak activity cluster for Right hand grasp overt/attempt movement activity at S1
Time Frame: Single visit
Population: Individuals with hand impairment due to cervical spinal cord injury
Measure: Mean (Full Range); unit: mm^3 (cubic millimeters)
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 5
mm^3 (cubic millimeters) | 2588.8 [1394 to 2799]

6. Primary Outcome: Peak Activity Volume: Left Ankle Overt/Attempt Movement Activity at M1 - ALS
Description: Volume of peak activity cluster in M1 during overt/attempted movement of left ankle
Time Frame: Single visit
Population: Impairment of at least one arm/hand as a result of cervical spinal cord injury
Measure: Mean (Full Range); unit: mm^3 (cubic millimeters)
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 3
mm^3 (cubic millimeters) | 437 [118 to 936]

7. Primary Outcome: Peak Activity Volume: Right Toe Overt/Attempt Movement Activity at M1 - ALS
Description: Volume of peak activity cluster in M1 during attempted movement of right toe by individuals with ALS
Time Frame: Single visit
Population: Impairment of at least one arm/hand as a result of cervical spinal cord injury or amyotrophic lateral sclerosis. The ALS diagnosis should be possible, probably, or definite ALS based on El Escorial criteria.
Measure: Mean (Full Range); unit: mm^3 (cubic millimeters)
Groups:
- Individuals With ALS: Individuals with hand impairment due to amyotrophic lateral sclerosis
Arm/Group | Individuals With ALS
Number analyzed (Participants) | 3
mm^3 (cubic millimeters) | 251.5 [152 to 351]

8. Primary Outcome: Peak Activity Volume: Right Hand Grasp Overt/Attempt Movement Activity at M1 - ALS
Description: Volume of peak activity cluster in M1 during attempted right hand grasp movement by individuals with ALS
Time Frame: Single visit
Population: as for outcome 7
Measure: Mean (Full Range); unit: mm^3 (cubic millimeters)
Arm/Group | Individuals With ALS
Number analyzed (Participants) | 3
mm^3 (cubic millimeters) | 238.5 [23 to 454]

9. Primary Outcome: Location of Peak Activity (X-coordinate) for Right D1 Attempt Movement - SCI
Description: This is the X-axis (right to left of head) coordinate for location of peak activity for attempted movement of right D1.
Time Frame: Single visit
Population: The x-axis coordinate is the left-to-right location of the peak activity.
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 5
mm | 176.4 [159 to 183]

10. Primary Outcome: Location of Peak Activity (Y-coordinate) for Right D1 Attempt Movement - SCI
Description: This is the Y-axis (vertical) coordinate for location of peak activity for attempted movement of right D1.
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 5
mm | 67 [61 to 79]

11. Primary Outcome: Location of Peak Activity (Z-coordinate) for Right D1 Attempt Movement - SCI
Description: This is the Z-axis (front to back of head) coordinate for location of peak activity for attempted movement of right D1.
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With Spinal Cord Injury
Number analyzed (Participants) | 5
mm | 103.2 [95 to 110]

12. Primary Outcome: Location of Peak Activity (X-coordinate) for Left Ankle Overt/Attempt Movement Activity - ALS
Description: This is the X-axis (right to left of head) coordinate for location of peak activity for M1 during overt/attempted movement of left ankle.
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With ALS
Number analyzed (Participants) | 3
mm | 123.33 [120 to 128]

13. Primary Outcome: Location of Peak Activity (Y-coordinate) for Left Ankle Overt/Attempt Movement Activity - ALS
Description: This is the Y-axis (right to left of head) coordinate for location of peak activity for M1 during overt/attempted movement of left ankle.
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With ALS
Number analyzed (Participants) | 3
mm | 63.67 [60 to 66]

14. Primary Outcome: Location of Peak Activity (Z-coordinate) for Left Ankle Overt/Attempt Movement Activity - ALS
Description: This is the Z-axis (right to left of head) coordinate for location of peak activity for M1 during overt/attempted movement of left ankle.
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With ALS
Number analyzed (Participants) | 3
mm | 87.67 [84 to 95]

15. Primary Outcome: Location of Peak Activity (X-axis): Right Hand Grasp - SCI
Description: Location of peak activity (X-axis coordinate): Right hand grasp overt/attempt movement activity at S1
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Groups:
- Individuals With SCI: Impairment of at least one arm/hand as a result of cervical spinal cord injury
Arm/Group | Individuals With SCI
Number analyzed (Participants) | 5
mm | 163.6 [153 to 176]

16. Primary Outcome: Location of Peak Activity (Y-axis): Right Hand Grasp - SCI
Description: Location of peak activity (Y-axis coordinate): Right hand grasp overt/attempt movement activity at S1
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With SCI
Number analyzed (Participants) | 5
mm | 59.4 [54 to 75]

17. Primary Outcome: Location of Peak Activity (Z-axis): Right Hand Grasp - SCI
Description: Location of peak activity (Z-axis coordinate): Right hand grasp overt/attempt movement activity at S1
Time Frame: Single visit
Measure: Mean (Full Range); unit: mm
Arm/Group | Individuals With SCI
Number analyzed (Participants) | 5
mm | 93 [86 to 105]

ADVERSE EVENTS:
Time Frame: 1 visit (approximately 4 hours)
Description: Adverse events are observed by the participant or the study team. These may include: falling during transfer to MRI surface, claustrophobia, burn from metal implant.
Groups:
- Participants With Spinal Cord Injury; Participants With Amyotrophic Lateral Sclerosis: Individuals will be asked to imagine movements or sensations while fMRI is used to measure brain activity.
  Motor or sensory imagery: Brain activity will be measured using fMRI while participants imagine different movements or sensations in order to assess the organization of sensorimotor cortical activity after injury.
Arm/Group | Participants With Spinal Cord Injury | Participants With Amyotrophic Lateral Sclerosis
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

LIMITATIONS AND CAVEATS:
Area of peak activity was not calculated and instead the volume and location coordinates were provided for peak activity of various movements associated with hand movements. Also, the volume or locations of activity that had statistically significant activity were included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT04723823/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT04723823/ICF_001.pdf